CLINICAL TRIAL: NCT01452412
Title: Placebo-controlled Randomized Clinical Trial of Alkali Therapy in Patients With Chronic Kidney Disease
Brief Title: Alkali Therapy in Chronic Kidney Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Michal L. Melamed, Associate Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-408; R01DK087783 (NIH)
Record Dates: First submitted 2011-10-12; First posted 2011-10-14 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Chronic Kidney Disease; Metabolic Acidosis
Keywords: Alkali; Sodium bicarbonate; Kidney disease; Acidosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acidosis; Kidney Diseases | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (2):
- Sodium bicarbonate (Experimental): 0.4 mEq/kg/day ideal body weight to be taken once a day
  Interventions: Drug: Sodium bicarbonate
- Placebo (Placebo Comparator): placebo dosage/frequency equivalent to sodium bicarbonate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium bicarbonate — 0.4 mEq/kg/day ideal body weight to be taken once a day
  Arms: Sodium bicarbonate
Drug: Placebo — To be taken on the same schedule as the active arm
  Arms: Placebo

SUMMARY:
Kidney disease is a common medical condition. Individuals with kidney disease develop a build-up of acid in their blood. This acid can affect their muscles, bones, glucose metabolism and kidneys. The investigators will test alkali treatment, to treat acid build-up, in a randomized placebo-controlled clinical trial to evaluate effects on muscles, bones, glucose metabolism and kidney.

ELIGIBILITY:
Inclusion Criteria:

* Estimate GFR <= 45 and >15 ml/min/1.73m2
* Age >18

Exclusion Criteria:

* Previous chronic treatment with alkali within the last 3 months (including sodium bicarbonate, calcium carbonate or baking soda)
* bicarbonate level <20 or >25 mEq/L
* New York Heart Association Class III or IV heart failure
* Systolic blood pressure >180 mmHg
* Initiation of ESRD treatment planned within 6 months
* Kidney transplantation
* Treatment with immunosuppressives within the last 3 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hostetter, MD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Derived] Brightwell CR, Kulkarni AS, Paredes W, Zhang K, Perkins JB, Gatlin KJ, Custodio M, Farooq H, Zaidi B, Pai R, Buttar RS, Tang Y, Melamed ML, Hostetter TH, Pessin JE, Hawkins M, Fry CS, Abramowitz MK. Muscle fibrosis and maladaptation occur progressively in CKD and are rescued by dialysis. JCI Insight. 2021 Dec 22;6(24):e150112. doi: 10.1172/jci.insight.150112. PMID 34784301
- [Derived] Melamed ML, Horwitz EJ, Dobre MA, Abramowitz MK, Zhang L, Lo Y, Mitch WE, Hostetter TH. Effects of Sodium Bicarbonate in CKD Stages 3 and 4: A Randomized, Placebo-Controlled, Multicenter Clinical Trial. Am J Kidney Dis. 2020 Feb;75(2):225-234. doi: 10.1053/j.ajkd.2019.07.016. Epub 2019 Nov 5. PMID 31699517

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Bicarbonate | Placebo
Started | 74 | 75
Completed | 46 | 58
Not Completed | 28 | 17
Not completed — Withdrawal by Subject | 15 | 11
Not completed — Adverse Event | 4 | 3
Not completed — Lost to Follow-up | 5 | 3
Not completed — Death | 1 | 0
Not completed — Initiated dialysis | 1 | 0
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Bicarbonate | Placebo | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (14.1) | 61.6 (10.9) | 61 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 42 | 80
  Male | 36 | 33 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 63 | 63 | 126
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 47 | 86
  White | 24 | 16 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 12 | 23
Serum bicarbonate [Mean (Standard Deviation); unit: mEq/L] | 24 (2.2) | 24.1 (2.6) | 24 (2.2)
estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: ml/min/1.73m2] | 36.2 (11.1) | 36.4 (11.4) | 36.3 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Sit to Stand to Sit Speed: Time Taken to Sit to Stand to Sit 10 Times
Description: Sit to stand to sit x10 speed (time to perform sit to stand to sit 10 times) will be measured and compared between groups.
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 74 | 75
seconds | 23.8 (5.8) | 22.9 (6.5)

2. Primary Outcome: DEXA of Wrist
Description: The investigators will evaluate changes in bone mineral density at the wrist.
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 74 | 75
g/cm2 | 0.75 (0.23) | 0.73 (0.17)

3. Secondary Outcome: Hand-grip Strength
Description: Hand-grip strength will be measured in all participants
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 74 | 75
kg | 27.3 (9.8) | 24.9 (10.2)

4. Secondary Outcome: Estimated GFR
Description: Estimated GFR
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 74 | 75
ml/min/1.73m2 | 38.5 (17.7) | 36.3 (14.5)

5. Secondary Outcome: Quality of Life - Physical Function Domain
Description: Short Form- 36 (SF-36) will be performed in all participants. We will evaluate effects on the Physical Function Domain. The Physical Function Domain is scored from 0 to 100 with higher scores meaning better physical functioning.
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 74 | 75
score on a scale | 40 (12) | 43 (11)

ADVERSE EVENTS:
Arm/Group | Sodium Bicarbonate | Placebo
All-Cause Mortality (participants affected / at risk) | 1/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 20/74 | 15/75
Other Adverse Events (participants affected / at risk) | 29/74 | 41/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Bicarbonate (N=74) | Placebo (N=75)
All-cause hospitalization (General disorders) | 20 (20) | 15 (15) — Hospitalizations were collected, not cause of hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Bicarbonate (N=74) | Placebo (N=75)
Serum bicarbonate >=30 (Renal and urinary disorders) | 9 (9) | 5 (5)
Serum bicarbonate <=18 (Renal and urinary disorders) | 2 (2) | 4 (4)
Serum potassium <=3.5 (Renal and urinary disorders) | 4 (4) | 2 (2)
Serum potassium >= 5.0 mEq/L (Renal and urinary disorders) | 14 (14) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No